## informed consent

Research Project Title: Clinical Implications of Internet + Wearable Devices in Multiple

Pre-Rehabilitation for Television-Assisted Thoracoscopic Surgery

Research Leader: Zijia Liu

Tel: 18511891786, 010-69152020

Research Organization: Peking Union Medical College Hospital, Chinese Academy of

Medical Sciences, Beijing, China

Please read this document carefully, all the information provided herein will help you whether or not to participate in the study. Research is voluntary and will not affect medical behavior. You need to understand the research risks, benefits, and alternatives.

1. purpose of the study:

Prehabilitation refers to the process of optimizing a patient's functional status through preoperative optimization to better tolerate surgical stress. Whether aerobic exercise prehabilitation strategies alone versus multiple prehabilitation strategies are beneficial in elderly patients undergoing thoracoscopic surgery needs to be proven.

- To assess the perioperative physical functional status of patients undergoing thoracoscopic surgery in elderly patients;
- To investigate whether giving outpatient anesthesia prehabilitation guidance earlier and performing ordinary multimodal home-based strategies or multimodal prehabilitation strategies assisted by "Internet + wearable devices" during the preoperative waiting period for elderly patients undergoing thoracoscopic surgery can improve the perioperative prognosis of the patients, and enable the patients to return to their daily life more quickly, daily life.

## 2. Content, methodology and procedures of the study:

## List of study times for all patients

| research period | 数据收集 |
|---|---|
| Initial outpatient | Collection of basic information, underlying medical history, |
| visit | contact information |
| | Basic quality of life and psychological assessment |
| • | Anesthesia risk assessment (including 6-minute walk test and |
| | baseline pulmonary function) |
| | Perioperative medication guidance |

| | Perioperative FAQs |
|---|---|
| The day before | Quality of Life and Psychological Assessment |
| surgery | Anesthesia Pre-Operative Assessment and Visits |
| First 3 days after | Assessment of short-term prognosis |
| surgery | |
| 4 weeks after | Perform psychological and midterm prognostic assessments |
| surgery | Outpatient follow-up |
| | • Measurement of 6-minute walk test |

Participating patients were randomly divided into two groups, namely, the multilink prehabilitation group and the "Internet + wearable device" group. Patients in both pre-rehabilitation groups implemented a home-based pre-rehabilitation program during the pre-operative phase until the day before surgery.

- 3. Possible risks and benefits of participating in the study. Risks: Any study should be considered a risk:
- Risks: any study has risks, and the main risk in this study comes from the potential inconvenience to patients during postoperative follow-up.

The preoperative anesthesia clinic assessment group alone was only accepted for more detailed assessment and follow-up; the two prehabilitation groups were safe and feasible interventions for teaching and advising on home prehabilitation strategies. There were no additional risks for patients in any of the three groups.

There were no additional medical costs associated with this study.

 Benefit: All patients may receive a more comprehensive preoperative anesthesia evaluation and more careful postoperative follow-up.

Patients in the prehabilitation group may have a faster recovery, with reduced length of stay and hospitalization costs.

- 4. Consultation about the content: You have the right to consult about the content of the study at 18511891786, 69152020 (investigator's phone number), and you have the right to consult about your rights or the related risks at 69154494 (Ethics Review Committee phone number).
- 5. Withdrawal from the study: Your participation in this study is completely voluntary. If, for any reason, you do not want to participate or continue to participate in this study, it will not affect your rights in any way. In addition, you may withdraw from this study at any time and for any reason without any loss to you. (You may also be asked to withdraw by your doctor or

the researcher if you do not follow your doctor's instructions or if your doctor wants you to do so for your health and well-being.)

- 6. Compensation for the study: If you suffer damage to your health as a result of participating in this study, you will be reimbursed by your health insurance in accordance with the rules and regulations, and Peking Union Medical College Hospital will not be responsible for any additional compensation.
- 7. Confidentiality: The medical information you obtain by participating in this study will be kept confidential. The results of the study will be published in academic journals without disclosing any personally identifiable information about you. Peking Union Medical College Hospital will keep all records of your participation in this study, as well as relevant hospital and office records, and no one will be allowed to access this information without authorization.
- 8. This informed consent form shall be executed in duplicate, one by the subject and one by the investigator, and shall be valid when signed by both parties.

## **Subject's Informed Consent:**

I have read and fully understand the above in detail and have given careful consideration to the above, particularly the rights, risks and benefits of my participation in this study. I volunteer to participate in this study and am willing to cooperate with the researchers. It is also declared that I may withdraw from this study at any time for any reason without loss of any legal rights.

| Subject's signature: | date: |
|------------------------------|-------|
| Signature of the researcher: | date: |